CLINICAL TRIAL: NCT01921907
Title: Phase 2 Double-blind, Randomized, Placebo-controlled, Parallel Group, Multi-center Study
Brief Title: Evaluation of a Topical Treatment for Actinic Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AD17137
Record Dates: First submitted 2013-07-31; First posted 2013-08-14 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-02

CONDITIONS: Actinic Keratosis of Face and Scalp
Keywords: Actinic keratosis; topical; dermatology; treatment; clinical study; double blinded
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Active (Experimental): topical treatment
  Interventions: Drug: AD17137 topical treatment
- Placebo (Placebo Comparator): topical treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AD17137 topical treatment
  Arms: Active
Drug: Placebo
  Arms: Placebo

SUMMARY:
A topical treatment applied twice daily for 4 weeks to induce disappearance of facial actinic keratosis (AK). First 4 weeks treatment (visit 1, 2 and 3 at 0,2 an 4 weeks) treated as a double blind parallel study. From weeks 4 to 7 (visit 3 to visit 4) all patients to be treated by the active component.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 30 to 90 years old, inclusive, in good general health
* Clinical diagnosis of Actinic Keratosis
* At least 2 clinically diagnosed, 3-15 mm AK lesions on face or scalp
* Patient is competent to understand and sign a consent form, and is willing and able to follow study procedures and attend all visits
* Female patients of childbearing potential must have a negative urine pregnancy test prior to receiving study medication
* Sexually active women of childbearing potential participating in the study must use a medically acceptable form of contraception
* Pharmacologic methods of contraception should be stable for 1 month prior to Visit 1 and be maintained at same dose during the study

Exclusion Criteria:

* Patients who had been treated with: 5-FU, diclofenac, retinoids, ingenol mebutate or imiquimod within 4 weeks of study, immunomodulators, or interferon/interferon inducers or systemic immunosuppressants within 8 weeks of study, cryodestruction, curettage, photodynamic therapy, surgical excision on the treatment area within 4 weeks of study, systemic cancer therapy, UVA therapy, UVB therapy, laser abrasion, dermabrasion
* History of hereditary angio-edema, Epilepsy or Parkinson's Disease
* Erythroderma or history of immunodeficiency disorders
* Pregnancy, lactation or patient who is not practicing effective contraception
* History of alcohol and drug abuse within 5 years of screening
* Known hypersensitivity or previous allergic reaction to any of the components of the study medication
* Having a member of the same household in the trial
* Patient has participated in an investigational clinical, surgical, drug or device study within the past 30 days
* Patients who in the opinion of the investigator should not be included in the study for any reason, including inability to follow procedures

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Complete Clearance (100% of AK lesions) from baseline (Visit 1) to Visits 3 and 4. Complete Clearance (100% of AK lesions) from baseline (Visit 1) to Visits 3 and 4. | baseline to Week 7

SECONDARY OUTCOMES:
Partial Clearance (75% of AK lesions) from baseline (Visit 1) to Visits 3 and 4. | baseline to Week 7
Mean change in lesion size | baseline to Week 7
Change in Investigator Global Assessment | baseline to Week 7
Mean change in lesion number | baseline to Week 7
Change in Patient Global Assessment | baseline to Week 7

CONTACTS AND LOCATIONS:
Locations (1):
- Maccabi Health Clinic, Tel Aviv, Tel Aviv, Israel